CLINICAL TRIAL: NCT01719718
Title: The Influence of Closing the Gap on Postoperative Seroma and Recurrences in Laparoscopic Ventral Hernia Repair.
Acronym: CLOSURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012/075
Record Dates: First submitted 2012-10-30; First posted 2012-11-01 (Estimated); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Ventral Hernia
Keywords: ventral hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Closure (Active Comparator)
  Interventions: Procedure: Closure of hernia defect.
- Non-Closure (Sham Comparator)
  Interventions: Procedure: No closure of the hernia defect.

INTERVENTIONS:
Procedure: Closure of hernia defect. — Laparoscopic ventral hernia repair with closure of the hernia defect (mesh augmentation technique).
  Arms: Closure
Procedure: No closure of the hernia defect. — Conventional laparoscopic ventral hernia repair without closure of the hernia defect (defect bridging technique).
  Arms: Non-Closure

SUMMARY:
A multicenter prospective randomized controlled trial comparing closure versus non-closure of the hernia defect between 2 and 5 cm in width using a tissue separating mesh (Physiomesh™) in laparoscopic ventral hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from the patient or his/her legal representative
* Ventral or incisional hernia requiring elective surgical repair
* Diameter between 2 and 5cm in width
* Midline and flank hernias are eligible

Exclusion Criteria:

* No written informed consent
* 'Hostile' abdomen, open abdomen treatment
* Contraindication to pneumoperitoneum
* Emergency surgery (incarcerated hernia)
* Parastomal hernia
* Subxiphoidal hernia
* Subcostal hernia
* Suprapubic hernia
* Clean-contaminated or contaminated field
* Hernia diameter >5cm in width
* Pregnancy
* Non-compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Seroma formation after 4 weeks. | 4 weeks after surgery.
  The seroma formation is checked by clinical evaluation.

SECONDARY OUTCOMES:
Pain, discomfort and esthetic evaluation after 4 weeks. | 4 weeks after surgery.
  Pain, discomfort and esthetic evaluation is performed after 4 weeks by clinical evaluation and the Visual Analogue Scale.
Pain, discomfort and esthetic evaluation after 1 year. | 1 year after surgery.
  Pain, discomfort and esthetic evaluation is performed after 1 year by clinical evaluation and the Visual Analogue Scale.
Pain, discomfort and esthetic evaluation after 2 years. | 2 years after surgery.
  Pain, discomfort and esthetic evaluation is performed after 2 years by clinical evaluation and the Visual Analogue Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Berrevoet, MD, PhD, FACS, Principal Investigator — University Hospital, Ghent
Locations (6):
- Belgium (6):
  - Algemeen Stedelijk Ziekenhuis, Aalst
  - Imelda Hospital, Bonheiden
  - St Vincentius Hospital, Deinze
  - Ghent University Hospital, Ghent
  - Maria Middelares, Ghent
  - Hôpital Mont Godinne, Namur

REFERENCES:
- See also: Related Info — http://www.uzgent.be